CLINICAL TRIAL: NCT01186562
Title: A Double-Blind, Randomized, Placebo Controlled Intervention Study to Assess the Impact of Sitagliptin 100 mg/Day for 1 Year on Insulin Independence Following Pancreatectomy and Autoislet Transplantation
Brief Title: Sitagliptin Therapy to Improve Outcomes After Islet Autotransplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1006M83756
Record Dates: First submitted 2010-08-04; First posted 2010-08-23 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Pancreatitis; Diabetes
Keywords: Pancreatitis; Pancreatectomy; Islet autotransplant; Sitagliptin; Diabetes
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg PO daily
  Arms: Sitagliptin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to test the effects of sitagliptin on the need for insulin (the hormone that lowers blood sugars) by patients who receive a pancreatectomy and islet autotransplant for chronic pancreatitis.

DETAILED DESCRIPTION:
At the current time, about one-third of patients are insulin independent (do not need to take insulin) after autotransplant, but the other two-thirds still need some insulin. Sitagliptin works by increasing the amount of a hormone called glucagon-like peptide 1, or GLP-1, in the body which then increases the amount of insulin that is made by the beta cells(the insulin producing cell of the islets). GLP-1 might also help protect beta cells from dying under stressful conditions and increase the production of new beta cells.

The primary goal of this study is to see if taking sitagliptin for one year after islet autotransplant increases the number of patients who achieve and maintain insulin independence. Other goals of this study are to see if sitagliptin reduces the amount of insulin injections needed or helps the islets make more insulin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for total pancreatectomy and IAT at UM

Exclusion Criteria:

* Pre-existing diabetes mellitus or hyperglycemia with fasting glucose ≥115 mg/dl
* Medical conditions which, in the opinion of the investigator, might impact islet function (e.g asthma or inflammatory disease requiring chronic systemic corticosteroids)
* Significant renal disease: serum creatinine levels of >3.0 mg/dL in men and >2.5 mg/dL in women, or end-stage renal disease requiring hemodialysis or peritoneal dialysis.
* For female subjects, plans to become pregnant or unwillingness to practice birth control for 18 months.
* Islet yield <1,000 IE/kg body weight (exclusion for treatment with drug/placebo)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-08; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melena Bellin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harindhanavudhi T, Yang Y, Hodges JS, Pruett TL, Kirchner V, Beilman GJ, Bellin MD. Body Composition is Associated With Islet Function After Pancreatectomy and Islet Autotransplantation for Pancreatitis. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e496-e506. doi: 10.1210/clinem/dgaa790. PMID 33124670

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 54 | 29
Completed | 50 | 27
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 54 | 29 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11) | 42.6 (10.3) | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 23 | 67
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 54 | 29 | 83

OUTCOME MEASURES:

1. Primary Outcome: Insulin Independence
Description: percentage of patients insulin independent
Time Frame: 12 months
Population: N's reflect patients that returned for study follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 50 | 29
percentage of participants | 42 | 45

2. Secondary Outcome: Insulin Independence
Description: percentage of patients insulin independent
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 50 | 27
percentage of participants | 36 | 44

3. Secondary Outcome: Area Under the Curve (AUC) C-peptide (ng/dL*Min)
Description: AUC C-peptide obtained from a mixed meal test (measured time 0 to 2 hours after Boost HP)
Time Frame: 12 months
Population: Patients with vomiting, NPO restrictions (due to chronic GI illness) were not able to complete MMTT. The N for each group reflects the number of patients who successfully completed this assessment.
Measure: Mean (Standard Error); unit: ng*min/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 48 | 27
ng*min/dL | 273 (20) | 273 (27)

4. Secondary Outcome: AUC C-peptide
Description: AUC C-peptide (ng/dL*min) from mixed meal tolerance test (measured times 0 to 2 hours after Boost HP)
Time Frame: 18 months
Population: Patients with vomiting, NPO (Nothing by Mouth) restrictions (due to chronic GI illness) were not able to complete MMTT. (Mixed meal Tolerance Test) The N for each group reflects the number of patients who successfully completed this assessment.
Measure: Mean (Standard Deviation); unit: min*ng/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 44 | 24
min*ng/dL | 274 (20) | 235 (27)

5. Secondary Outcome: Acute C-peptide Response (ACR) to Glucose
Description: Derived from intravenous gluocose tolerance testing (0 to 10 minute measures after dextrose bolus)
Time Frame: 12 months
Population: This test required two IVs. In patients for whom 2 IVs could not be placed successfully, this test could not be performed. N's reflect number of patients completing this test.
Measure: Mean (Standard Error); unit: min*ng/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 49 | 26
min*ng/dL | 9.9 (1.2) | 7.2 (1.6)

6. Secondary Outcome: Acute C-peptide Response (ACR) to Glucose
Description: Derived from intravenous glucose tolerance test (0 to 10 minute measures after IV dextrose bolus)
Time Frame: 18 months
Population: as for outcome 5
Measure: Mean (Standard Error); unit: min*ng/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 46 | 23
min*ng/dL | 6.9 (1.0) | 6.0 (1.4)

ADVERSE EVENTS:
Time Frame: 18 months
Description: from treatment start to 18 month follow up
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 31/54 | 26/29
Other Adverse Events (participants affected / at risk) | 54/54 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=54) | Placebo (N=29)
AST Metabolic/Laboratory (Metabolism and nutrition disorders) | 1 | 0
Abdomen Pain (Gastrointestinal disorders) | 8 | 6
Appendicitis Infection (Infections and infestations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Biliary Tree Infection (Gastrointestinal disorders) | 1 | 1
Blood Infection (Infections and infestations) | 0 | 1
Catheter Infection (Infections and infestations) | 0 | 1
Cellulitis Infection (Infections and infestations) | 2 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Constipation Gastrointestinal (Gastrointestinal disorders) | 3 | 3
Dehydration Gastrointestinal (Gastrointestinal disorders) | 5 | 2
Diabetes Type 1 Endocrine (Endocrine disorders) | 0 | 1
Diarrhea Gastrointestinal (Gastrointestinal disorders) | 2 | 2
Dizziness Neurology (Nervous system disorders) | 0 | 1
Edema Limb Lymphatics (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue Constitutional Symptoms (General disorders) | 1 | 0
Fever Constitutional Symptoms (Infections and infestations) | 7 | 3
Fracture Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 | 1
GI Hemorrhage/Bleeding (Gastrointestinal disorders) | 1 | 0
Headache Pain (Nervous system disorders) | 0 | 1
Hyperglycemia Metabolic/Laboratory (Endocrine disorders) | 0 | 1
Hypoglycemia Metabolic/Laboratory (Endocrine disorders) | 1 | 3
Kidney Infection (Infections and infestations) | 1 | 0
Nausea Gastrointestinal (Gastrointestinal disorders) | 1 | 2
Obstruction Gastrointestinal (Gastrointestinal disorders) | 0 | 1
Obstruction Bowel Gastrointestinal (Gastrointestinal disorders) | 7 | 5
Opioid Withdrawl Pain (General disorders) | 1 | 0
Other- J tube Malfunction Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Other- Maligancy Gastrointestinal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Other-Suicide attempt (Psychiatric disorders) | 0 | 1
Pain Gastrointestinal (Gastrointestinal disorders) | 0 | 1
Penicillin Allergy/Immunology (Immune system disorders) | 1 | 0
Perihepatic abscess Infection (Infections and infestations) | 0 | 1
Peritoneal Cavity Infection (Infections and infestations) | 1 | 0
Pleural Effusion Pulmonary/ Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia Infection (Infections and infestations) | 1 | 0
Syncope Neurology (Nervous system disorders) | 1 | 0
Thrombosis Vascular (Blood and lymphatic system disorders) | 1 | 0
Ulcer Jejunum Gastrointestinal (Gastrointestinal disorders) | 0 | 1
Ulcer: duod. Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Vomiting Gastrointestinal (Gastrointestinal disorders) | 5 | 0
Weight Loss Constitutional Symptoms (General disorders) | 0 | 1
Wound Infection (Infections and infestations) | 4 | 0
Wound complication Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Wound- Hernia Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=54) | Placebo (N=29)
ALT Metabolic/Laboratory (Metabolism and nutrition disorders) | 6 | 4
AST Metabolic/Laboratory (Metabolism and nutrition disorders) | 8 | 3
Abdomen Pain (Gastrointestinal disorders) | 13 | 9
Abdomen_infection Infection (Infections and infestations) | 0 | 1
Achy Constitutional Symptoms (General disorders) | 1 | 0
Acne Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Albumin low Metabolic/Laboratory (Metabolism and nutrition disorders) | 25 | 14
Alk Phos high Metabolic/Laboratory (Metabolism and nutrition disorders) | 3 | 0
Alkalosis (metabolic) Metabolic/Laboratory (Metabolism and nutrition disorders) | 1 | 0
Allergic Rhinitis Allergy/Immunology (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anal Fissure Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Anorexia Gastrointestinal (Gastrointestinal disorders) | 1 | 1
Anxiety Neurology (Psychiatric disorders) | 1 | 1
Arthritis Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 | 2
Ascites Gastrointestinal (Gastrointestinal disorders) | 5 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Biliary Tree Leak Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Bladder Infection (Infections and infestations) | 1 | 0
Blood Infection (Infections and infestations) | 1 | 0
Blurred Vision Ocular/ Visual (Eye disorders) | 1 | 0
Bronchitis Infection (Infections and infestations) | 1 | 1
Bronchospasm Pulmonary/ Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catheter Infection (Infections and infestations) | 1 | 0
Cellulitis Infection (Infections and infestations) | 4 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest/ Throat NOS Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colitis Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Concussion Neurology (Nervous system disorders) | 0 | 1
Confusion Neurology (Nervous system disorders) | 3 | 0
Constipation Gastrointestinal (Gastrointestinal disorders) | 7 | 3
Cough Pulmonary/ Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Creatinine Metabolic/Laboratory (Metabolism and nutrition disorders) | 0 | 1
Cyst Removal Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 | 1
Dehydration Gastrointestinal (Gastrointestinal disorders) | 2 | 1
Dental- Tooth Infection (Infections and infestations) | 2 | 1
Depression Neurology (Nervous system disorders) | 1 | 1
Diarrhea Gastrointestinal (Gastrointestinal disorders) | 17 | 10
Distention Gastrointestinal (Gastrointestinal disorders) | 0 | 1
Dizziness Neurology (Nervous system disorders) | 1 | 2
Dry Eye Syndrome Ocular/ Visual (Eye disorders) | 1 | 0
Dry Mouth Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Edema Limb Lymphatics (Musculoskeletal and connective tissue disorders) | 9 | 4
Elevated WBC Blood/BoneMarrow (Blood and lymphatic system disorders) | 1 | 1
Extremity Pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Fatigue Constitutional Symptoms (General disorders) | 6 | 0
Fever Constitutional Symptoms (Infections and infestations) | 6 | 7
Flu-like syndrome Syndromes (Infections and infestations) | 8 | 6
Fracture Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 0 | 2
GERD Gastrointestinal (Gastrointestinal disorders) | 1 | 0
GI Hemorrhage/Bleeding (Gastrointestinal disorders) | 2 | 0
Headache Ocular/ Visual (Nervous system disorders) | 1 | 0
Headache Pain (Nervous system disorders) | 13 | 7
Hematoma Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1 | 2
Hemoglobin Blood/BoneMarrow (Blood and lymphatic system disorders) | 27 | 13
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hot Flashes Endocrine (Endocrine disorders) | 1 | 0
Hyopalbuminemia Metabolic/Laboratory (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia Endocrine (Endocrine disorders) | 1 | 0
Hypoglycemia Metabolic/Laboratory (Endocrine disorders) | 0 | 1
Hypokalemia Metabolic/Laboratory (Metabolism and nutrition disorders) | 1 | 0
Hypotension Caridac General (Cardiac disorders) | 0 | 1
Hypothyroidism Endocrine (Endocrine disorders) | 1 | 0
INR Coagulation (Blood and lymphatic system disorders) | 1 | 0
Ileus Gastrointestinal (Gastrointestinal disorders) | 1 | 0
Insomnia Constitutional Symptoms (Nervous system disorders) | 3 | 0
Irregular Menses Sexual/ Reproductive Function (Endocrine disorders) | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Kidney Infection (Infections and infestations) | 2 | 0
Kidney Pain (Renal and urinary disorders) | 1 | 0
Libido Sexual/ Reproductive Function (Reproductive system and breast disorders) | 1 | 0
Liver Infection (Gastrointestinal disorders) | 0 | 1
Memory Impairment Neurology (Nervous system disorders) | 1 | 0
Middle Ear Infection (Infections and infestations) | 1 | 1
Middle Ear Pain (Ear and labyrinth disorders) | 1 | 0
Mood Alteration-Panic attack (Psychiatric disorders) | 0 | 1
Mood Alteratons: Anxiety (Psychiatric disorders) | 2 | 0
Mood alteration other (Psychiatric disorders) | 1 | 0
Mood alteration-Depression (Psychiatric disorders) | 0 | 1
Muscle Cramps Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Spasm Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea Gastrointestinal (Gastrointestinal disorders) | 17 | 6
Neuropathy Sensory Neurology (Nervous system disorders) | 0 | 1
Neuropathy/Sensory Neurology (Nervous system disorders) | 1 | 0
Other- Eye Swelling Allergy/Immunology (Eye disorders) | 0 | 1
Other- Kidney Stone Renal/ Genitourinary (Renal and urinary disorders) | 2 | 1
Other- Ovarian cyst Sexual/ Reproductive Function (Reproductive system and breast disorders) | 1 | 0
Other- eye redness/ lid swelling Ocular/ Visual (Eye disorders) | 1 | 0
Other-Congestion Pulmonary/ Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Other-Meningioma Neurology (Nervous system disorders) | 1 | 0
Other/ Temp Intol Constitutional Symptoms (Gastrointestinal disorders) | 1 | 0
PTT Coagulation (Blood and lymphatic system disorders) | 1 | 0
Peritoneal Cavity Infection (Infections and infestations) | 1 | 1
Pharynx Infection (Infections and infestations) | 4 | 0
Photophobia Ocular/ Visual (Eye disorders) | 1 | 0
Platelets Blood/BoneMarrow (Blood and lymphatic system disorders) | 0 | 1
Pneumonia Infection (Infections and infestations) | 1 | 2
Psychosis Neurology (Psychiatric disorders) | 3 | 1
Pulmonary/Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash Dermatology/Skin (Skin and subcutaneous tissue disorders) | 4 | 5
Rhinitis Allergy/Immunology (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Seizure Neurology (Nervous system disorders) | 1 | 0
Shingles Infection (Infections and infestations) | 1 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus Infection (Infections and infestations) | 6 | 2
Syncope Neurology (Nervous system disorders) | 1 | 0
Throat Pain (Gastrointestinal disorders) | 7 | 2
Thrombosis Vascular (Blood and lymphatic system disorders) | 1 | 3
Tinnitus Auditory/Ear (Ear and labyrinth disorders) | 1 | 0
Toe Infection (Infections and infestations) | 1 | 0
Tonsilitis Infection (Infections and infestations) | 1 | 0
Tooth Pain (Gastrointestinal disorders) | 0 | 1
Triglyceride serum high Metabolic/Laboratory (Metabolism and nutrition disorders) | 0 | 2
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 4
Vagina Infection (Infections and infestations) | 1 | 0
Vision Blurred Vision Ocular/ Visual (Eye disorders) | 1 | 0
Voice Change Pulmonary/ Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Vomiting Gastrointestinal (Gastrointestinal disorders) | 11 | 7
Vomitting Gastrointestinal (Gastrointestinal disorders) | 0 | 1
Weakness Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Weight Gain Constitutional Symptoms (General disorders) | 15 | 4
Weight Loss Constitutional Symptoms (General disorders) | 25 | 17
Wound Infection (Skin and subcutaneous tissue disorders) | 0 | 1
Wound complication Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
It is also possible that the study is not powered enough to detect small differences in insulin independence. The feasibility of conducting any larger trial in the small population of adult islet autograft recipients is limited, however.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No